CLINICAL TRIAL: NCT01874158
Title: DNA Clearance of Uncomplicated Trichomonas Vaginalis Infections in HIV Negative Women
Status: Completed | Type: Observational
Sponsor: Tulane University Health Sciences Center (Other)
Collaborators: Louisiana State University Health Sciences Center in New Orleans (Other)
Responsible Party: Principal Investigator, Patricia Kissinger, Professor, Tulane University Health Sciences Center
Organization: Tulane University (Other)
Other Study IDs: 8115
Record Dates: First submitted 2013-06-06; First posted 2013-06-10 (Estimated); Last update posted 2016-12-19 (Estimated); Status verified 2016-12

CONDITIONS: Trichomonas Vaginitis
Keywords: Trichomonas vaginalis
MeSH Terms: conditions — Trichomonas Vaginitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 1 vaginal swab collected at screening for In-pouch 3 vaginal swabs collected at enrollment, PCR, gram stain, and future microbiome study At each of 3 follow-up visits, 3 vaginal swabs, PCR, In-pouch, and future microbiome study At the 4th follow-up visit, 4 vaginal swabs, PCR, In-pouch, gram stain, and future microbiome study.
  All swabs, except at screening, are self-collected.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- TV postive women: All women who are TV positive by wet prep or in-pouch and meet the inclusion exclusion requirements.

SUMMARY:
The objective of this study is to screen treated Trichomonas vaginalis (TV) positive women weekly using culture and Polymerase Chain Reaction (PCR) to determine how long TV DNA is detectable post treatment and to examine potential confounders to clearance such as bacterial vaginosis.

DETAILED DESCRIPTION:
Trichomonas vaginalis (TV), the most common sexually transmitted infection in the world, is associated with inflammation of the vagina, cervix, and urethra; low birth weight; preterm delivery; pelvic inflammatory disease; and may increase the risk of acquiring and transmitting genital herpes and HIV. Repeat infections are common, ranging from 5% - 31%, and have similar health outcomes as primary infections. Given the high prevalence of TV, the absence of a national screening program, the deleterious reproductive outcomes associated with TV and the potential for a TV infection to increase HIV transmission, reducing repeat TV infections is an important targeted public health approach. However, rescreening for TV should not happen until there is sufficient time for the parasites and DNA to clear from the vaginal cavity after treatment. HIV negative women who attend Delgado Personal Health Center will be asked to enroll in the screening component in order to test them for TV using InPouch culture along with the standard TV screening of wet preparation. The objective of this study is to screen treated TV positive women weekly using culture and Polymerase Chain Reaction to determine how long TV DNA is detectable post treatment and to examine potential confounders to clearance such as bacterial vaginosis. The outcome of interest will be a negative PCR result indicating that TV DNA has cleared.

ELIGIBILITY:
Inclusion Criteria:

* English speaking females
* >18 years old
* HIV-negative
* a patient at the Delgado Personal Health Center

Exclusion Criteria:

* HIV+ women

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: English speaking HIV- women over the age of 18 who are TV positive
Sampling Method: Non-Probability Sample
Enrollment: 99 (Actual)
Dates: Start 2012-11; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
TV negative by PCR, post treatment | 4 weeks
  Women are assessed for TV at each weekly visit by PCR. They are considered cleared of the remnant DNA after PCR is negative.

CONTACTS AND LOCATIONS:
Overall Officials: Patricia J Kissinger, PhD, Principal Investigator — Tulane University School of Public Health and Tropical Medicine
Locations (1):
- Delgado Personal Health Center, New Orleans, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No